# **Informed Consent**

| Screening Number: | |
|-----------------------------|----------------|
| Random Number: | |
| Sponsor: Plastic Surgery, X | ijing Hospital |

**Version Number: 2.0** 

Version Date: Dec 08, 2017

### **Project name:**

Comparative study on the clinical efficacy of golden microneedles and 1565nm non-ablative lattice laser in the treatment of eyelid pouches

#### Possible benefits of participating in the study:

Benefits to the subject: improvement of eyelid pouch, skin texture, skin relaxation, etc. Benefits for social groups: Evaluation of safety and effectiveness of non-invasive treatment for patients with BLEs.

### Possible risks Complications and preventive treatment:

| Possible risks | Prevention and treatment |
|---|---|
| BLEs asymmetry | Bilateral treatment plan interchanged 3 times, followed up for 4 weeks |
| | and 12 weeks; severe cases of surgery pain |
| Pain | Local 5% compound lidocaine cream film sealed surface anesthesia, if |
| | necessary neurological stagnation |
| Swelling, Bruising | Cold pack for 30 minutes before and after treatment. Keep the head |
| | high for at least 3 days after treatment. |
| Exudation,punctate | Compression to reduce bleeding, external medical repair accessories to |
| hemorrhage | promote skin repair, reduce exudation. |
| Pigment changes | Apply broad-spectrum sunscreen if necessary oraling VC, VE ect. |

## Who should I contact if I have questions or difficulties?

If you have any questions about this study, or if you have any discomfort during the study, you can always contact your research doctor: Name: Wenjie Dou . Phone: +86\_182\_0926\_1917\_Address: Plastic Surgery, Xijing Hospital\_.

If you have any questions about your rights as a research subject, please contact:

Ethics Committee of Xijing Hospital, Tel: 029-84771794.

## **Informed Consent Statement Subject**

#### **Informed Consent Statement:**

The research physician has informed me of the research background, purpose, procedures, risks, and benefits of this study, and I have also read the written information. I have read this informed consent and agree to participate in this study. I have also been told who to contact when I have questions or want further information. I understand that I can withdraw from the study at any time and that my future treatment will not be affected by this. By signing this informed consent, I agree that my physiological and demographic data can be used under the conditions described in this informed consent. I agree that this informed consent form will be made in duplicate, signed by me and the research doctor, and both parties will keep one copy.

| Subject name: | <u> </u> |
|--------------------|-----------------|
| Subject signature: | (block letters) |
| Date of signature: | |

#### **Research doctor's notification statement:**

I have informed the subject "Gold microneedles and 1565nm non-ablative "Comparison of the clinical efficacy of sexual lattice laser in the treatment of blepharoplasty", the research background, purpose, steps, risks and benefits of the project, giving him / her enough time to read the informed consent, discuss with others, and answer its related questions

Questions from the study; I have informed the subject of their contact information when they encounter a problem; I have informed the subject that they can withdraw from the study at any time during the study without any reason.

| Research doctor's name: | <u> </u> |
|------------------------------|-----------------|
| Research doctor's signature: | (block letters) |
| Signature date: | |